CLINICAL TRIAL: NCT00676988
Title: A Cross Sectional Study To Determine The Relationship Between Serum Infliximab Concentration And Efficacy In Patients With Luminal Crohn's Disease
Brief Title: Study to Determine Relationship Between Serum Infliximab and Efficacy in Luminal Crohn's Disease Patients
Acronym: X-Sectional
Status: Completed | Type: Observational
Sponsor: University of Western Ontario, Canada (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Other Study IDs: RP0701
Record Dates: First submitted 2008-05-08; First posted 2008-05-13 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Crohn's Disease
Keywords: Luminal Crohn's Disease; Infliximab
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum infliximab concentrations and CRP levels.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observation: Subjects with Luminal Crohn's Disease receiving infliximab

SUMMARY:
To assess the relationship between the change in Crohn's Disease Activity Index (CDAI) scores and trough serum infliximab concentration in subjects who are scheduled to receive infliximab infusions at an interval of 8 weeks.

DETAILED DESCRIPTION:
This cross sectional study will evaluate a sample of 360 subjects with luminal Crohn's disease who are receiving infliximab in 15-20 Canadian infusion centres. The sample will be stratified by disease activity [mild = CDAI <150, moderate/severe = CDAI ≥150] and whether or not subjects are on concomitant immunosuppressive therapy. Thus 4 strata will be created consisting of 90 subjects each. Consent will be obtained prior to or at Visit 1, subjects will retrospectively complete a CDAI diary card for the preceding 7 days and blood work will be drawn prior to infliximab infusion. Four weeks thereafter at Visit 2, subjects will provide an additional blood sample to measure serum infliximab concentrations and CRP levels. Between Visits 1 and 3, subjects will complete daily CDAI diary entries. Visit 3 will take place at the next scheduled infusion, 8 weeks after Visit 1 (+/- 7 days ).

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (18 years of age or older at time of consent)
* Confirmed diagnosis of inflammatory luminal Crohn's Disease
* Receive infliximab therapy and have received a minimum of 5 consecutive infusions at prescribed intervals (minimum of 24 weeks and maximum of 156 weeks on infliximab therapy)
* Plan to receive the next 2 infliximab infusions at 8-weekly intervals (+/- 7 days)
* Able to provide written consent

Exclusion Criteria:

* Active draining fistulizing Crohn's Disease
* Presence of an ostomy
* Diagnosis of ulcerative colitis
* Infliximab dose of >5mg/kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with Luminal Crohn's disease receiving infliximab at Canadian Infusion Centres
Sampling Method: Non-Probability Sample
Enrollment: 327 (Actual)
Dates: Start 2008-05; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian G Feagan, MD, Principal Investigator — Director Clinical Trials; Gordon R Greenberg, MD, Principal Investigator — co-principal investigator
Locations (2):
- Canada (2):
  - MedEmerg Infusion Clinics, Mississauga, Ontario
  - CIM - Centre d'Intervention Medicales Inc., Pointe-Claire, Quebec

REFERENCES:
- [Derived] Levesque BG, Greenberg GR, Zou G, Sandborn WJ, Singh S, Hauenstein S, Ohrmund L, Wong CJ, Stitt LW, Shackelton LM, King D, Lockton S, Ducharme J, Feagan BG. A prospective cohort study to determine the relationship between serum infliximab concentration and efficacy in patients with luminal Crohn's disease. Aliment Pharmacol Ther. 2014 May;39(10):1126-35. doi: 10.1111/apt.12733. Epub 2014 Apr 1. PMID 24689499